CLINICAL TRIAL: NCT02906982
Title: A Randomized Trial Evaluating the Efficacy of a Gum Health Formulation on Teeth Whitening in Patients With Gingivitis and Periodontitis
Brief Title: Evaluating the Efficacy of a Gum Health Formulation on Teeth Whitening in Patients With Gingivitis and Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glo Science, Inc. (Industry)
Collaborators: EEC Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLO-001
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Tooth Discoloration; Periodontal Diseases
Keywords: Periodontal diseases; Periodontitis; Gingivitis; Teeth Whitening; Dental Plaque Index; Periodontal Index; Teeth Whitening Agents; Tooth Discoloration; Mean Probing Depth; Pocket Depth
MeSH Terms: conditions — Tooth Discoloration; Periodontal Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gum health formulation in intra-oral device (Experimental): The interventional gum health formulation is applied to the participant's mouth by means of an intra-oral device for a single eight-minute application, daily. Participants instructed to brush their teeth with a toothbrush and toothpaste twice daily, morning and night.
  Interventions: Other: Gum health formulation in intra-oral device
- Gum health formulation on toothbrush (Experimental): The interventional gum health formulation is applied to the participant's mouth by means of a toothbrush and toothpaste, plus the gum health formulation, for two-minute applications, twice daily, morning and night.
  Interventions: Other: Gum health formulation on toothbrush
- Control group (split-mouth design) (No Intervention): The control group did not receive the interventional gum health formulation. Participants instructed to brush their teeth with a toothbrush and toothpaste twice daily, morning and night. In addition, participants instructed to floss only half of their mouth daily, and the non-flossed half serves as the untreated comparative control receiving no intervention.

INTERVENTIONS:
Other: Gum health formulation in intra-oral device — The intervention is a gum health formulation for periodontal disease care and teeth whitening to be used within an accelerating intra-oral device.
  Other Names: ECO Balance; GLO Science intra-oral accelerating device
  Arms: Gum health formulation in intra-oral device
Other: Gum health formulation on toothbrush — The intervention is a gum health formulation for periodontal care and teeth whitening to be used on a toothbrush alongside standard toothpaste.
  Other Names: ECO Balance
  Arms: Gum health formulation on toothbrush

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel gum health formulation, when used in an intra-oral device or on a toothbrush, for teeth whitening and clinical improvements in periodontal diseases.

DETAILED DESCRIPTION:
Over half of the American population suffers from some form of periodontal disease, while millions of Americans are electing for teeth whitening procedures every year. The study is designed to assess the efficacy of a novel gum health formulation on teeth whitening in the context of gingival inflammation. Further, the study aims to assess the efficacy of the novel gum health formulation as an adjunct to the current standard of care in the treatment of gingivitis and periodontitis, depending on the severity of disease. As the dental professional community is whitening teeth in an environment of gingival inflammation, a single product that whitens teeth and controls inflammation is a novel treatment approach and highly desirable among patients and consumers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, understand and sign an Informed Consent form
* Good general health as evidenced by the medical history
* Between 18 and 65 years of age
* A minimum of 20 teeth, excluding crowns and third molar teeth
* A mean whole mouth Gingival Index score of >2.0 at baseline
* Sites with <7mm pocket depth
* Willing to abstain from all oral hygiene procedures for 12-18 hours prior to clinical visits
* Willing to abstain from eating and drinking in the morning of visits, only drinking water
* Willing to abstain from chewing gums, oral whitening products, mouthwashes and tobacco products for the study duration
* Ability to understand and follow study protocol
* No known history of allergy to dairy products or their ingredients, relevant to any ingredient in the test products

Exclusion Criteria:

* Chronic use of photosensitizing medications including NSAIDs, antidepressants, antibiotics and beta blockers
* Diagnosis of diabetes mellitus
* Presence of orthodontic appliances
* Presence of large restorations
* Crown or veneer at the anterior of both upper and lower teeth (including premolar teeth)
* A soft or hard tissue tumor of the oral cavity
* Carious lesions
* Severe internal (tetracycline stains) and external discolouration (fluorosis)
* Diagnosis of severe chronic periodontitis, aggressive periodontitis, acute necrotizing ulcerative gingivitis or generalized gingival recession >2mm as evidenced by clinical oral exam
* Participating in another clinical trial or oral product study
* Pregnant or breast-feeding women
* Allergy to home bleaching products such as hydrogen peroxide and carbamide peroxide
* Use of antibiotics within 3 months of enrolment
* History of drug use that is associated with gum overgrowth (i.e., Dilantin, nifedipine, etc.)
* Chronic use of medication such as steroids, anti-coagulant medications, immunosuppressant medications or any other medications or medical conditions that in the opinion of the investigator would interfere with the evaluation or confound interpretation of the study results
* Medical condition which requires pre-medication prior to dental visits/procedures
* Smokers
* Patients who have received quadrant or maintenance scaling & root planing and/or periodontal surgical therapy within 6 months prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Tooth Shade Value over 45 Days | Baseline, Day 14, Day 28, Day 45
  Tooth Shade Value was measured using a Vita Shade Guide and the measurement was transformed to a standardized value.

SECONDARY OUTCOMES:
Plaque Index | Baseline, Day 14, Day 28, Day 45
  Periodontal probe will be swept along the buccal and lingual surfaces and plaque is noted.
Gingival Index | Baseline, Day 14, Day 28, Day 45
  Periodontal probe will be placed under the gingival margin and swept along the buccal and lingual surfaces and bleeding is noted.
Bleeding Index | Baseline, Day 14, Day 28, Day 45
  Bleeding will be assessed after probing. A dichotomous scoring system is used at six sites per tooth using one and zero for presence or absence, respectively.
Mean Probing Depth | Baseline, Day 14, Day 28, Day 45
  Pocket depth will be determined with a UNC-15 periodontal probe at six sites per tooth rounded to the next lower whole millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Edgard El Chaar, DDS, MS, Principal Investigator — EEC Institute, Inc.
Locations (1):
- EEC Institute, Inc., New York, New York, United States